CLINICAL TRIAL: NCT02797834
Title: Isolation and Characterization of the Extracellular Vesicles Secreted by the Human Endometrium to the Endometrial Fluid
Brief Title: Isolation and Characterization of the Extracellular Vesicles Secreted by the Human Endometrium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Felip Vilella, Research Director, Igenomix
Other Study IDs: 1603-IGX-017-FV
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Extracellular Vesicles
Keywords: Extracellular vesicles; Endometrial fluid; Menstrual cycle; Exosomes; Microvesicles; Apoptotic bodies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, proteins, lipids and other metabolits will be analyzed in the different samples of the endometrial fluid.
  These samples will be completely exhausted during the analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Endometrial Fluid: Endometrial fluid samples from healthy and fertile women in their natural cycles, with ages ranging from 18 to 35 years, normal karyotype, negative for HIV, HBV, HCV and RPR, BMI ranging from 18 to 30 Kg/m2 (both included) and regular menstrual cycle (3-4/28-30 days).
  This unique assignment group will be divided into 5 subgroups attending to the moment of the menstrual cycle in which the patient could be classified: phase I (days 0-8), phase II (days 9-14), phase III (days 15-18), phase IV (days 19-24) and phase V (days 25-30).
  Interventions: Procedure: Endometrial fluid collection

INTERVENTIONS:
Procedure: Endometrial fluid collection

SUMMARY:
The main aim of this study is to describe the morphology, size distributions and specific markers of the different vesicles populations present in the human endometrial fluid. To further characterize the vesicles populations, contents of these membrane compartments (i.e.: DNA, RNA, proteins, lipids and other small metabolites) will be assessed by using mass spectrometry and next generation sequencing techniques. The objective here is to relate a specific vesicles composition to the moment of the cycle, to a normal physiological endometrial function and to the transmission of functionalities from the mother to the embryo.

DETAILED DESCRIPTION:
In the last decades, the emission of membrane enclosed compartments, more commonly regarded as extracellular vesicles, has been established as a new mechanism of communication either between cells of a complex organism, between unicellular organisms or between unicellular organism and host. These vesicles have been described in all body fluids and are currently classified into three types according to the mechanism by which they are formed: exosomes, with sizes ranging from 30 to 150 nm (formed intracellularly); microvesicles, between 100 and 1000 nm (formed from the cell membrane) and apoptotic bodies, with sizes greater than 1 µm (produced by cells undergoing programmed cell death).

Endometrial fluid is a viscous liquid present in the uterine cavity originating from the different cell types that form the uterus and serum exudates. It offers a precise view of the context in which the embryo implants and can be retrieved by a minimally invasive technique.

The main objective of this pilot study is to isolate and characterize the extracellular vesicles secreted by the endometrium to the endometrial fluid, being this the first time that this fact is being described. It is intended to standardize a method for the isolation of the different vesicles populations present within the endometrial fluid (i.e.: apoptotic bodies, microvesicles and exosomes), based on serial differential centrifugations and filtration. Morphological characterization of the isolated vesicles will be done at three levels: study of the external morphology by transmission electron microscopy, characterization of the different vesicles populations surface markers by Western Blot and analysis of the vesicles populations size distributions by Nanoparticle Tracking Analysis.

The second part of the study is directed to assess the content of the extracellular vesicles throughout the menstrual cycle. For this purpose, a canonical menstrual cycle of 28 to 30 days has been classified in 5 phases: phase I (days 0-8), phase II (days 9-14), phase III (days 15-18), phase IV (days 19-24) and phase V (25 to 30). The experimental design for vesicles contents description consists of two levels of comparison: (1) analysis of differential contents of the different populations of vesicles in the same phase of the menstrual cycle and for each of the phases and (2) analysis of differential contents of the same population of vesicles in each phase of the cycle and for each of the vesicular populations. This characterization of the vesicular contents will be made using mass spectrometry techniques to analyze the protein, lipid and other small metabolites composition. Their presence aims to be related both to the moment of the cycle and to a normal physiological function of the endometrium. On the other hand, analysis of DNA and RNA contents of these vesicular populations by massive sequencing will be performed. The objective here is to analyze the transmission of functionalities to target cells as well as the potential predictive usefulness of these molecules to determine the moment of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women in natural cycles.
* Age: 18 to 35 years (both included).
* Normal karyotype.
* Negative serological results for HIV, HBV, HBC, RPR.
* BMI: 18-30 Kg/m2 (both included).
* Regular menstrual cycle (3-4/28-30 days).

Exclusion Criteria:

* Patients who had carried a IUD device in the previous 3 months.
* Patients who had taken hormonal contraceptives in the previous 2 months.
* Adnexal or uterine pathologies.
* Polycystic ovary syndrome.
* Patients suffering from serious or uncontrolled bacterial, fungal or viral infectious diseases that could potentially interfere with the participation of the patient or with the results of the study (evaluated by the principal researcher of the research team).
* Any unstable disease or medical condition that could interfere with the study or put in risk the health of the patient (evaluated by the principal researcher of the research team).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Analysis in this study will be done using endometrial fluid samples retrieved from healthy, fertile, normal-cycling women which meet the inclusion/exclusion criteria.
  These patients will be recruited in a single national centre: IVI Valencia. Their recruitment will be done during the routine clinical practice by the research group in the previously mentioned centre.
  The research group will be in charge of checking patients' medical reports and getting in contact with those patients that meet the selection criteria and are willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Morphological characterization of the extracellular vesicles | 3 months
  Assessment of the morphology of the extracellular vesicles using transmision electron microscopy by either ultrathin cuts and positive staining or deposition and positive staining techniques.
  The aim is to differentiate between vesicle populations thanks to their external aspects and size.
Size distribution profiles characterization of the extracellular vesicles | 45 days
  Analysis of the size distribution of the vesicles contained in the different extracellular vesicles populations by using two Nanoparticle Tracking Analysis techniques: ZetaSizer Nano and NanoSight300.
  The expected outcome is a set of graphs with size range data of the vesicles in the different populations and vesicle concentration data when using NanoSight300.
Characterization of extracellular vesicles populations by specific markers | 45 days
  Analysis of population-specific markers by Western Blot in order to further differentiate endometrial fluid vesicles populations.
  The aim is to differentiate populations based on the presence or absence of these markers.

SECONDARY OUTCOMES:
Qualitative (names) and quantitative (expression levels) information about the different biomolecules that could be present in the samples: DNA, RNA, proteins, lipids and other small metabolites. | three years

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Vilella, BSc PhD, Principal Investigator — Igenomix
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No